CLINICAL TRIAL: NCT05583994
Title: OPTIM-PARK II -A New Intervention for Optimisation of Community Resources and Systems of Support to Enhance the Process of Living With Parkinson's Disease: a Feasibility Trial
Brief Title: Optimising Community Resources and Support to Enhance Living With Parkinson's Disease
Acronym: OPTIM-PARKII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Solent NHS Trust (Other Government); Salisbury NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 308776
Record Dates: First submitted 2022-09-01; First posted 2022-10-18 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: community; Parkinson's Disease; Carers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Control and intervention groups (usual care vs new intervention)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants cannot be blinded to the intervention they are receiving. Outcome assessors and the main investigators are blinded to group allocation and will not have access to the intervention treatment lists. Only the statistician performing the randomization, the team member supporting the coordinator and the coordinator who is delivering the intervention are aware of group allocation.
  However, previous experience has shown that participants may occasionally and inadvertently inform assessors of the treatment they are receiving. The research team aim to reduce this effect by explicit reminders to participants before assessment visits. The research team shall ask all assessors to record their estimate of which group they think the participant belongs, and their confidence in that prediction. This will enable to test whether inadvertent loss of blinding leads to bias, and to adjust for any bias detected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care ( control) (No Intervention): All participants in the trial will continue with their usual care as deemed appropriate by health care providers, this will usually comprise attendance at medical clinics, medication, and visits from PD nurse specialists. Participants may attend group activities or access resources as part of their usual care, though from experience such sessions are rarely intensive or prolonged. Participants will be asked to record their usual care and encouraged to avoid changing that practice unless specifically requested by a health care worker during the time they are participating in the trial.
- Optim Park Intervention (Experimental): A central component of the Optim-Park II intervention is to offer a single point of contact with a coordinator (appointed for the purpose of delivering the Optim-Park II intervention) to assess participants needs, have a discussion with participants to identify 3 main problems/targets PwPD and carers would most like to address based on their needs and then link up and refer participants to available community resources.
  The coordinators will deliver the Optim-Park intervention for PwPD and their carers in three consultations: a consultation after the baseline assessment and randomization has been undertaken at the point of "entrance" to the study; a consultation in the middle of this period; and a follow-up consultation at "exit" at 3 months. Each consultation can last between 30 min and up to 2 hours. Each consultation can be with the pair of PwPD and carer or if appropriate, separately.
  Interventions: Other: Optim Park Intervention

INTERVENTIONS:
Other: Optim Park Intervention — For participants receiving the Optim-Park II intervention, the aim is to enhance the process of living with Parkinson's Disease for the person with PD and the family-carer by building a multisectoral care pathway, with a special focus on how to optimize the use of resources and systems of support in the community in disadvantaged populations in UK.
  Arms: Optim Park Intervention

SUMMARY:
This is a multi-centre, single-blinded, randomized, controlled trial for PwPD (people with Parkinson's Disease) to compare (i) OPTIM-PARK II (a novel personalized treatment based on the latest published research evidence and results from our extensive development work undertaken in OPTIM-PARK I) and routine care with (ii) routine care alone. The research team will provide a personalized list of available resources to the routine care arm at the end of the trial. The trial aims to recruit 60 PwPD and their carers (n=60) in the UK. This trial took place in 4 countries (Denmark, Norway, Spain and UK) but only Spain and UK included control groups, data collection in these two countries started in October 2022, after the iterative phase of the trial.

At the screening visit participants will be asked whether they would also be willing to take part in an additional qualitative study. A subgroup of participants will be selected from those that have indicated a willingness to take part in the qualitative study. Also, at the screening visit participants will be asked whether they have a carer. Having a carer is not a pre-requisite for PwPD being recruited into the trial. It is likely that some PwPD in the trial may not have a suitable carer. Where one is available, they will be invited to join the trial: if there is more than one, the main family carer, as identified by the PwPD, will be approached.

DETAILED DESCRIPTION:
This is a multi-centre, single-blinded, randomised, controlled trial for PwPD to compare (i) OPTIM-PARK II (a novel personalised treatment based on the latest published research evidence and results from our extensive development work undertaken in OPTIM-PARK I) and routine care with (ii) routine care alone. The research team will provide a personalised list of available resources to the routine care arm at the end of the trial. The trial aims to recruit 60 PwPD and their carers (n=60) in the UK. This trial took place in 4 countries (Denmark, Norway, Spain and UK) but only Spain and UK included control groups, data collection in these two countries started in October 2022, after the iterative phase of the trial.

Participants allocated to the control group will received usual care and participants in the intervention group the Optim Park intervention.

This intervention will consist of the following:

First consultation with PwPD and carer "entrance" at point of entry to the study

The initial consultation with the PwPD and the carer will be a face-to-face consultation in the participants own home or at the clinic/primary care centre/community hub based on participants preference.

This consultation will include steps which are detailed below.

Step 1. Welcome and clarification of expectations PwPD and their carer will be welcomed to the Optim-Park II intervention. In this step, the coordinator and the PwPD and the carer will get to know each other and the clarification of expectations for this intervention will take place. The coordinator will outline that the consultation is intended to allow participants to gain information about available public and private services, community and volunteer-based resources that are available to them. In this step, the coordinator will record the resources that the PwPD and carer have already accessed or used in the past and will record this in the resource log.

Step 2. Personalised assessment and needs clarification A personalised assessment will be carried out with PwPD and carers in collaboration with the coordinator to explore and identify their needs.

For PwPD To enable this process, the PwPD and the coordinator will have access to the Living with long term conditions scale (completed during the baseline assessment) which they can use as a conversation starter to encourage PwPD to reflect on their experience of living with PD. The coordinator might also use the map of resources for clarification of needs.

For carers The carer and the coordinator will have access use the Carer Support Needs Assessment Tool (CSNAT) (completed during the baseline assessment) which they can use as a conversation starter to explore in which areas the carer require support to enable them to care for the PwPD and to preserve their own health and well-being within their caregiving role. The coordinator might also use the map of resources for clarification of needs.

Step 3. Choice of focus Based on the personalised assessment and needs clarification the coordinator, in collaboration with the PwPD and the carer, will identify the main 3 issues/areas they each want to address or need the most help and support. The coordinator will document each of their 3 issues using the Log of resources. This way the coordinators and PwPD and the carer can revisit this in the following consultations.

Step 4. Information selection Together the coordinator, PwPD and carer will decide about what resources would like to be informed about or referred to in order to tackle the main issues/areas identified in Step 2. The coordinator will in collaboration with the PwPD and carer identify which resources could best address accommodate their issues/areas of focus. Together the coordinator, the PwPD and the carer will select resources from the map of resources that are considered appropriate and acceptable for the PwPD and the carer. The coordinator will use the Log of resources to help the PwPD and the carer identify and record what were chosen to be most beneficial to their current situation and according to their expressed needs.

Step 5. Enable use of resources The coordinator will inform the PwPD and their carer about the resources and professional services available that they have selected in the previous step, and about how to access those resources/services. The coordinator will provide clear and concise information and not use technical language and outline potential individual benefits that the PwPD and carer could achieve and how this might support addressing the problems identified in step 2.

The Coordinator will use the Map of Resources to inform the PwPD and carer of the resource options available in their area. The information provided by the Coordinator may be complemented with the delivery of printed or digital material (eg: web pages; and a copy of the Map of Resources in a version designed for PwPD and carer).

The Coordinator will use the Log to record the information they have provided to PwPD and carer about community resources and professional services.

The main objective of this step is that PwPD and carers are informed so that they can use the resources as and when they want to access them. In addition, referrals, signposting and first contact can also be made in this step based on the personalized assessment of needs.

Step 6. Intervention Follow-ups The Coordinator in collaboration with PwPD and carers can decide and make the next appointment depending on when and how the next follow-up consultation will take place. It is recommended to specify the day, time and place of the next consultation before ending the initial consultation. The PwPD and their carer will be informed that they can contact the coordinator with any problems and queries via phone or email at any point without having to make another appointment.

Second consultation: Intervention "as needed" This second consultation will be initiated by the coordinator if they have not heard back from the PwPD by phone in the middle of the 3-month follow-up.

The coordinator will ask the PwPD and carer about any thoughts and progress made or problems encountered following their discussion in the previous consultation. In particular, the coordinator might ask about the three problems identified in the initial consultation and doubts or uncertainties that have arisen after their initial consultation.

If the PwPD and carer have not found the identified resources useful or helpful, the coordinator will offer to inform them of other or different resources. If the PwPD or carer are struggling to make the first contact or engaging with available resources, the coordinator will offer to support the participants. At the end of this phone call consultation, the coordinator in collaboration with PwPD and carers will decide on the date, place and time of the next and last consultation.

Third consultation: Intervention exit This third and final consultation will be face-to-face in the participants own home or at the clinic/primary care centre, by phone or digital, based on participant preference 3 months after entry to the intervention.

The coordinator will ask the PwPD and Carer about their progress made in dealing with the main 3 problems identified during the initial consultations. The coordinator will record which resources were accessed, continued or discontinued and record how useful participants found these resources in relation to addressing the main 3 problems identified.

At the end of the meeting, the coordinator will answer any final questions and ensure that participants have a copy of the map of local resources.

ELIGIBILITY:
Inclusion Criteria:

* PwPD are eligible to be included in the trial if they meet the following criteria:

  1. Have a confirmed Consultant's diagnosis of Parkinson's disease.
  2. Live at home.
  3. Able to give informed consent.
  4. Able to understand and follow commands.
  5. Willing to take part in the Optim Park II intervention.

Carers of PwPD are eligible to be included in the trial if they meet the following criteria:

1. The PwPD they are caring for has given informed consent.
2. Live at home.
3. Able to give informed consent.
4. Able to understand and follow commands.
5. Willing to take part in the Optim Park II intervention.

Exclusion Criteria:

* Participants who are currently hospitalised or acutely unwell will not be eligible to being included in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Resources used in the community (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Resources identified and used as recorded in the Resource log (by the coordinator) and in the resource log diary (by patients and carers)

SECONDARY OUTCOMES:
Parkinson Disease Quality of Life 39 questionnaire (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Quality of Life Person with Parkinson Disease (0-100) (lower scores better Quality of Life)
Parkinson Disease quality of life Carer Scale (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Quality of Life Carer (0-100) (lower scores better Quality of Life)
Caregiver Burden Scale (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Caregiver Burden (0-84) (higher scores indicate more burden)
Duke University of Carolina Social support Questionnaire (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Social support (1-5 average score) (higher scores meaning better social support)
Health and social care resource use sheet (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Economic analysis
Euro Quality of Life 5 Dimension (assessing change) | Completed at baseline and 3 months post randomisation follow-up assessment
  Economic analysis (1-15 individual questions (1 best posible score) and Visual Analogue Scale (0-100, 100 best health possible)

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (2):
  - Hospital Universitario la Princesa, Madrid, Spain, Madrid
  - Autonomous University of Madrid/Nursing Department, Madrid
- United Kingdom (2):
  - Salisbury NHS Foundation Trust, Salisbury, Hampshire
  - University of Southampton, Southampton, Hampshire